CLINICAL TRIAL: NCT06085560
Title: Choice, Implementation Intentions and Colorectal Cancer Screening
Brief Title: Choose It and Use It: Choice, Implementation Intentions and At-Home Colorectal Cancer Screening
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Todd Lucas, C.S. Mott Endowed Professor, Michigan State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: 00007344
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Screening; Colorectal Cancer; Colonoscopy; FIT Kit; sDNA Kit; Cancer Screening; Health Communication; Health Disparities
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Design is factorial. After watching a brief didactic video, participants who opt to partake in colorectal cancer screening self select one of three screening modalities (colonoscopy vs. FIT Kit vs. sDNA Kit). Participants are then randomly assigned to one of three study arms (usual care vs. implementation intentions intervention vs. culturally targeted implementation intentions intervention). Screening selection and study arms are fully crossed.
Who Masked: Participant
Masking Description: Participants will be unaware of their assignment to usual care vs. intervention conditions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care Message (Active Comparator): Participants selecting a colorectal cancer screening will receive "usual care" from the FQHC.
  Interventions: Behavioral: Usual Care Message
- Implementation Intention Intervention: Standard Message (Active Comparator): Participants selecting a colorectal cancer screening will receive implementation intention messages in addition to the "usual care" from the FQHC.
  Interventions: Behavioral: Implementation Intention Intervention: Standard Message
- Implementation Intention Intervention: Culturally-Targeted Message (Experimental): Participants selecting a colorectal cancer screening will receive culturally-targeted implementation intention messages in addition to the "usual care" from the FQHC.
  Interventions: Behavioral: Implementation Intention Intervention: Culturally-Targeted Message

INTERVENTIONS:
Behavioral: Usual Care Message — Usual care is provided by the FQHC for the screening option chosen.
  Arms: Usual Care Message
Behavioral: Implementation Intention Intervention: Standard Message — Implementation Intention Intervention module includes standard messaging in addition to the usual care provided by the FQHC for the screening option chosen.
  Arms: Implementation Intention Intervention: Standard Message
Behavioral: Implementation Intention Intervention: Culturally-Targeted Message — Implementation Intention Intervention module includes culturally-targeted framing of health information messages in addition to the usual care provided by the FQHC for the screening option chosen.
  Arms: Implementation Intention Intervention: Culturally-Targeted Message

SUMMARY:
The goal of this study is to improve use of colorectal cancer screening among screening eligible African Americans who are served by Federally Qualified Health Centers in Michigan. The main questions it aims to answer are:

* To what extent to individual prefer and select to complete screening with colonoscopy versus stool-based (FIT Kit or sDNA) options?
* Can full completion of (i.e. follow-through with) screening with a selected modality be enhanced by delivery of a culturally targeted intervention?

Participants will learn about colonoscopy, FIT Kit and sDNA as recommended and widely used screening options. Participants will select a modality to complete their own screening with. Participants will then be randomized to one of three arms (usual care, standard intervention, culturally targeted intervention). Researchers will compare the extent to which intervention arms enhance completion rates across each of the three screening modalities.

DETAILED DESCRIPTION:
Background: African-Americans are more likely than other racial groups to develop and die from colorectal cancer (CRC). These disparities are largely due to lower rates of CRC detection among African-Americans. At-home CRC screening using a recommended screening tool - including fecal immunochemical testing (FIT Kit) and stool DNA testing (sDNA) ¬- could aid in reducing disparities. Yet, at-home screening remains underutilized, and little is known about preferences for specific at-home screening alternatives, despite that options present tradeoffs that likely influence uptake. Another challenge, including among African Americans, is that at-home screening suffers from low conversion - full completion of screening by individuals who are issued at-home screening kits. Implementation intentions may be an effective psychological tool for overcoming low conversion among African Americans.

Objective/Hypothesis: This study proposes to evaluate preference for and conversion rates associated with colonoscopy, FIT Kit and sDNA testing among low income Africans Americans, and will evaluate use of implementation intentions to promote uptake and conversion across these screening modalities.

Specific Aims: (1) To identify and compare preferences for colonoscopy versus annual FIT KIT testing versus stool DNA testing once every three years in a community sample of CRC screening-eligible African-Americans; (2) To identify and compare conversion of at-home CRC screening over three years among participants who elect to complete FIT Kit versus stool DNA testing for at-home CRC screening; (3) To determine the effectiveness of utilizing culturally targeted Implementation Intentions to promote conversion of colonoscopy and at-home CRC screening in screening eligible African-Americans.

Study design: In collaboration with clinical and community experts, the investigators will develop video materials to educate CRC screening eligible individuals about colonoscopy FIT Kit and sDNA as options for at-home CRC screening. In partnership with two Federally Qualified Health Center - one in Detroit, MI and one in Flint, MI - the investigators will provide access to these screening options and evaluate preferences for and conversion associated with each screening modality in a sample of screening eligible low-income African Americans. To consider strategies for enhancing conversion, the investigators will also evaluate a culturally-targeted approach to implementation intentions for use with CRC screening.

ELIGIBILITY:
Inclusion Criteria:

* African American, ages 45-72, Medicaid or Medicare insurance, enrolled in a FQHC, eligible for CRC screening (Colonoscopy more than 10 years ago, Sigmoidoscopy more than 5 years ago, FOB test more than 1 year ago, FIT kit more than 1 year ago, sDNA test more than 3 years ago, Never been screened).

Exclusion Criteria:

* All who do not meet inclusion criteria.

Ages: 45 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Colorectal Cancer Screening Modality Request Rates | up to 2 weeks
  Frequency (percentage) with which colonoscopy versus FIT Kit versus sDNA kit versus no screening are selected.
Colorectal Cancer Screening Completion Rate | up to 6 months
  Frequency (percentage of time) that chosen screening method is fully completed.
Theory of Planned Behavior Colorectal Cancer Screening Outcomes | collected immediately, up to 1 hour
  Self-report measures of colorectal cancer screening attitudes, norms, perceived control, intentions to be screened are each adapted from published research (Lucas et al., 2021). These items are constructed following recommended procedures to ensure construct validity and adequate behavioral specificity (Fishbein & Ajzen, 2011). All items use Likert-type scales that range from 1 (strongly agree) to 7 (strongly disagree).
Anticipatory Racism | collected immediately, up to 1 hour
  Adapted from published research (Lucas et al., 2021), all participants respond to questions that asked whether they believe racism would impact the benefits they could experience from obtaining colorectal cancer screening. Participants will then respond to three questions that ask, "In some way, my obtaining CRC screening would be impacted by racism," "Racism would undermine the value of CRC screening for me." and "Racism would negatively impact the accuracy of my CRC screening. Responses are collected using a 7-point Likert-type scale that ranged from 1 (strongly agree) to 7 (strongly disagree).

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available per requirements and sharing structures established by the American Cancer Society.
Supporting Information: Study Protocol
Time Frame: Upon Study Completion